CLINICAL TRIAL: NCT02247427
Title: Midterm Clinical Outcomes Related to Cardiac Resynchronization Therapy Deactivation of Super Responders
Brief Title: Clinical Outcomes Related to Cardiac Resynchronization Therapy Deactivation of Super Responders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yuksek Ihtisas Hospital (Other)
Responsible Party: Principal Investigator, Serkan Cay, Associate Professor, Yuksek Ihtisas Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: TYIH-132
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Cardiomyopathy
Keywords: Heart failure; Super responder
MeSH Terms: conditions — Cardiomyopathies; Heart Failure | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Off-pace group (Experimental): Deactivated device group
  Interventions: Device: Cardiac Resynchronization Therapy Device
- On-Pace group (No Intervention): Ongoing device activity group

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Device — Cardiac Resynchronization Therapy Device pacing activity, on or off
  Arms: Off-pace group

SUMMARY:
The purpose of this study is to determine clinical outcomes related to deactivation of Cardiac Resynchronization Therapy device in subjects with super response.

ELIGIBILITY:
Inclusion Criteria:

* super response to Cardiac Resynchronization Therapy
* near normal Left ventricular ejection fraction
* >99% pacing

Exclusion Criteria:

* <99% pacing
* atrial fibrillation
* ischemic cardiomyopathy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Clinical/Echocardiographic outcome | 12 months
  Clinical/Echocardiographic outcome including New York Heart Association class, 6-min walk test, Left ventricular ejection fraction, Left ventricular end- diastolic diameter, Left ventricular end-systolic volume, and Left ventricular end-systolic diameter.

SECONDARY OUTCOMES:
Mortality | 12 months
  Number of participants experiencing mortality
Heart failure hospitalization | 12 months
  Number of participants experiencing heart failure hospitalization
Cardiac Resynchronization Therapy Device intervention | 12 months
  Heart failure hospitalization Cardiac Resynchronization Therapy Device intervention for detected episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Cay, MD, Principal Investigator — Yuksek Ihtisas Hospital